CLINICAL TRIAL: NCT05067075
Title: Role of Continuous Glucose Monitoring Systems (CGMS) for Intrapartum Metabolic Control in Gestational Diabetic (GDM)Women
Brief Title: The CGMS in GDM Labor and Delivery Study
Acronym: CGMSGDMLABOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Woman's (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RP-21-017
Record Dates: First submitted 2021-09-22; First posted 2021-10-05 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy
Keywords: continuous glucose monitoring; labor; post-delivery

STUDY DESIGN:
Intervention Model Description: Blinded continuous glucose monitor will be compared with routine blood glucose monitoring
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Blinded CGM (Experimental): Blinded continuous glucose monitor Dexcom G6Pro
  Interventions: Device: Blinded CGM

INTERVENTIONS:
Device: Blinded CGM — CGM that records blood glucose but is not visible to patient or provider in real-time
  Other Names: Dexcom G6 Pro

SUMMARY:
Glucose control during labor is important for both fetus and mother. During labor and delivery, the goal is to maintain the sugars in the normal range as safely as possible as increased blood sugars 4-6 h prior to delivery leads to increased rates of hypoglycemia in the neonate. Neonatal hypoglycemia is a risk for the offspring of pregnant women with diabetes and occurs when fetal pancreatic hyperplasia is acutely stimulated by a high fetal glucose level derived from maternal hyperglycemia during labor. The maternal blood glucose level during delivery is a predictor of the neonatal blood glucose level. Modern continuous glucose monitoring (CGM) systems can capture the direction and magnitude of short-lived changes in interstitial glucose levels and are therefore useful for assessing glucose variability more accurately than self-monitoring blood glucose (SMBG) measurements. Indeed, it has already been demonstrated that intermittent blood glucose monitoring underestimates the number of hyperglycemic events, because blood glucose excursions can peak at different times of day. CGMs can help identify glycemic patterns in pregnancy, obtain and maintain glucose targets, and reduce hypoglycemia. Strict glycemic control during labor and delivery may reduce the risk of neonatal hypoglycemia. Two groups have reported on the use of CGM in type 1 diabetics during labor in small pilot studies. Another study looked at effects of maternal glucose levels in insulin-treated women during labor and delivery (2 to 8 h before birth) and resultant neonatal hypoglycemia. The researchers found that maternal hyperglycemia before delivery was correlated with neonatal hypoglycemia. Although more studies are needed, CGM use has promise as a therapy to improve outcomes in pregnancies associated with diabetes. In this study, the investigators plan to explore whether the use of blinded glucose monitoring during labor, delivery, and early postpartum supplementary to normally monitored plasma glucose measurements in women with gestational diabetes (GDM) would provide useful information to improve glycemia during labor in this diabetic population. All CGM data will be masked and therefore not available to participants, clinicians, or researchers at the time of delivery. Participants otherwise will receive standard clinical care. The blinded glucose monitoring data on glycemia throughout labor and post-delivery will be retrospectively assessed.

DETAILED DESCRIPTION:
Planning management for a diabetic parturient during labor and delivery is particularly challenging because of the demands of labor, dietary restrictions, and potential for operative delivery. The main goals can be summarized as: ensuring the avoidance of maternal hypoglycemia or hyperglycemia (which can increase the risk of neonatal hypoglycemia), ensuring the safe use of measures to manage glycemic control, and the provision of effective analgesia for labor. Currently available international guidelines for the peripartum management of pregnant women with diabetes focus on rigorous intrapartum glycemic control. Maternal hyperglycemia in women with pregestational and gestational diabetes mellitus can cause hypoglycemia in the neonate following delivery. In women with diabetes, maternal hyperglycemia leads to hyperplasia of pancreatic β cells in the fetus and an increase in fetal insulin concentrations. When the continuous supply of glucose is stopped after delivery, the neonate is at risk of developing hypoglycemia, which if untreated can have serious neurological consequences. The increase in fetal insulin also contributes to the excess growth of the fetus in mothers with hyperglycemia. Avoiding intrapartum maternal hyperglycemia may prevent fetal hyperglycemia and reduce the likelihood of subsequent neonatal hypoglycemia. A further potential concern relates directly to the woman. Immediately after delivery, postpartum insulin requirements decrease dramatically as a result of the rapid decrease in diabetogenic placental hormone levels and resulting dissipation of pregnancy-induced insulin resistance. Pregnant women with diabetes may be at greater risk of hypoglycemic episodes because awareness of the symptoms of hypoglycemia is reduced, and this is further exacerbated by tight glycemic control .

Glucose control during labor is important for both fetus and mother. During labor and delivery, the goal is to maintain the sugars in the normal range as safely as possible as increased blood sugars 4-6 h prior to delivery leads to increased rates of hypoglycemia in the neonate. Neonatal hypoglycemia is a risk for the offspring of pregnant women with diabetes and occurs when fetal pancreatic hyperplasia is acutely stimulated by a high fetal glucose level derived from maternal hyperglycemia during labor. The maternal blood glucose level during delivery is a predictor of the neonatal blood glucose level, and a high blood glucose level in the mother is associated with neonatal hypoglycemia. Continuous glucose monitoring (CGM) use appears to be safe and effective in pregnancies complicated by diabetes. Modern CGM systems can capture the direction and magnitude of short-lived changes in interstitial glucose levels and are therefore useful for assessing glucose variability more accurately than self-monitoring blood glucose (SMBG) measurements. Indeed, it has already been demonstrated that intermittent blood glucose monitoring underestimates the number of hyperglycemic events because blood glucose excursions can peak at different times of day. CGMs can help identify glycemic patterns in pregnancy, obtain and maintain glucose targets, and reduce hypoglycemia. CGM helps with treatment adjustments in pregnancies associated with diabetes. Strict glycemic control during labor and delivery may reduce the risk of neonatal hypoglycemia. In principle, "real-time" CGM might allow more rapid adjustment of insulin dosing and, thereby, yield better glycemic control than is possible with intermittent glucose monitoring. Two groups have reported on the use of CGM during labor in small pilot studies. Stenninger et al. reported that CGM was well tolerated in their 15 subjects and that elevated maternal glucose levels in the last 2 hours before delivery correlated with the need for intravenous glucose in the newborn. They found that multiple glycemic indices correlated positively with the need for neonatal intravenous glucose infusions. Iafusco et al. used real-time CGM in 14 subjects to guide insulin therapy during labor and found no cases of neonatal hypoglycemia. Another study looked at effects of maternal glucose levels in insulin-treated women during labor and delivery (2 to 8 hours before birth) and resultant neonatal hypoglycemia. In the this study, 45% (27/60) of women in the CGM group were compared with 100% (59/59) in the control group. Among women in the CGM arm, 10 infants developed hypoglycemia compared with 27 in the non-CGM group (37% vs. 46%, respectively; P = 0.45). The researchers found that maternal hyperglycemia before delivery was correlated with neonatal hypoglycemia.

Although more studies are needed, CGM use has promise as a therapy to improve outcomes in pregnancies associated with diabetes. In this study, the investigators plan to explore whether the use of blinded glucose monitoring during labor, delivery, and early postpartum supplementary to normally monitored plasma glucose measurements in women with gestational diabetes (GDM) would provide useful information to improve glycemia during labor in this diabetic population.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* a positive oral glucose tolerance test
* written informed consent
* labor scheduled for term induction (37-40 weeks)

Exclusion Criteria:

* prior diagnosis of type 1 or type 2 diabetes mellitus
* presence of infection
* Presence of significant systemic disease or other severe metabolic, endocrine, or medical co-morbidities
* History of bariatric surgery or other surgeries that induce malabsorption
* Long-term use (>2 weeks) of systemic steroids prior to enrollment
* Multiple pregnancy
* Participants already using glucose lowering medications (metformin or insulin) for diabetes before study entry (can be used after diagnosis of GDM)
* Fetal growth restriction due to placental dysfunction or known congenital anomaly
* History of major depressive or other severe psychiatric disorders or inpatient psychiatric treatment up to 1 year before enrolment
* Inability or refusal to comply with protocol

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — participant must be pregnant and have gestational diabetes during current pregnancy
Enrollment: 61 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Average percentage time in target glucose range | up to 10 days
  average time in hours and minutes spent in target glucose range

SECONDARY OUTCOMES:
average time spent in hyperglycemia (time above target range) | up to 10 days
  average time in hours and minutes spent with elevated blood sugar
average time spent in hypoglycemia (time below target range) | up to 10 days
  average time in hours and minutes spent with low blood sugar
neonatal hypoglycemia | up to 2 hours post delivery
  Neonatal hypoglycemia is defined as a 2-hour plasma glucose value < 2.1 mmol/l (47 mg/dL taken 2 hours after delivery

OTHER OUTCOMES:
postpartum 2 hour 75 gram OGTT results from mother | from 6 to 12 weeks after delivery
  glucose and insulin results from post delivery OGTT

CONTACTS AND LOCATIONS:
Overall Officials: Karen Elkind-Hirsch, PhD, Principal Investigator — Woman's Hospital, Louisiana
Locations (1):
- Woman's Hospital, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
The proposed research will involve a small sample (less than 65 subjects) recruited from clinical facilities at Woman's Hospital. Despite the removal of all identifiers, we believe that it would be difficult if not impossible to protect the identities of subjects. So even though the final dataset will be stripped of identifiers prior to release for sharing, we assume that there remains the possibility of deductive disclosure of subjects with unusual characteristics. Thus, we will make the de- identified data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed